CLINICAL TRIAL: NCT06270199
Title: Clinical Trial to Stablish the Security of Using Allogeneic Fetal Stem Mesenchymal Cells From Umbilical Cord, Expanded in Pre-term Patients Suffering of Bronchopulmonary Dysplasia.
Brief Title: Use of Mesenchymal Stem Cells in Pre-term Patients With Bronchopulmonary Dysplasia.
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PULMESCELL-2
Record Dates: First submitted 2024-01-16; First posted 2024-02-21 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary dysplasia; Preterm newbnorn; Mesenchymal stem cells
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Intervention Model Description: Parallel Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (Active Comparator): Standard cell therapy (control group)
  Interventions: Biological: Control
- Allogenic fetal mesenchymal stem cells from umbilical cord - three infusions (Experimental): Treatment: three infusions of MSC 5x10^6/Kg
  Interventions: Biological: Allogenic fetal mesenchymal stem cells from umbilical cord - three infusions
- Allogenic fetal mesenchymal stem cells from umbilical cord - six infusions (Experimental): Treatment: six infusions of MSC 5x10^6/Kg
  Interventions: Biological: Allogenic fetal mesenchymal stem cells from umbilical cord - six infusions

INTERVENTIONS:
Biological: Control — Standard treatment
  Arms: Control
Biological: Allogenic fetal mesenchymal stem cells from umbilical cord - three infusions — 3 doses of 5 million MSC will be administered
  Arms: Allogenic fetal mesenchymal stem cells from umbilical cord - three infusions
Biological: Allogenic fetal mesenchymal stem cells from umbilical cord - six infusions — 6 doses of 5 million MSC will be administered
  Arms: Allogenic fetal mesenchymal stem cells from umbilical cord - six infusions

SUMMARY:
Bronchopulmonary dysplasia (BPD) is a disease that affects preterm newborn patients, preventing their lungs from developing properly. Allogeneic fetal stem mesenchymal cells from umbilical cord could reduce the prevalence of BPD in this patients.

DETAILED DESCRIPTION:
Bronchopulmonary dysplasia (BPD) is a disease that affects preterm newborn patients, preventing their lungs from developing properly, and it is a disease that is nowadays increasing due to the improvement in the survival of this patients (affecting 15-50% of them).

In the Fase I Clinical Trial, the use of allogeneic fetal stem mesenchymal cells from umbilical cord proved to be safe, with no mortality or Adverse Events reported. The Fase II Clinical Trial is based in the hypothesis that the administation of mesenchymal stem cells is not only safe but feasible and can help reducing the chance of a preterm newborn patient developing BPD.

ELIGIBILITY:
Inclusion Criteria:

* Alive newborns weighing ≤ 1250 grams and GA ≤ 28 weeks, who are on mechanical ventilation with a FiO2 ≥0.3 between days 5 and 14 of life, with no immediate extubation foreseeable.

Exclusion Criteria:

* Presence of another concomitant congenital pathology at the time of inclusion: pulmonary malformations with compromised pulmonary function, active pulmonary haemorrhage, severe pulmonary hypoplasia, renal malformations with systemic compromise, congenital heart disease, polymalformative syndromes, chromosomopathies.
* Presence of refractory haemodynamic instability of any cause at the time of inclusion.
* Presence of severe neurological damage at the time of inclusion (HIV grade III or higher).
* Patients who have required major surgery in the 72 hours prior to inclusion.
* Patients who have necrotising enterocolitis (NEC) grades ≥II at the time of inclusion, according to the Bell classification.
* Patients who are children of a mother with HIV

Ages: 1 Month to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 75 (Estimated)
Dates: Start 2024-01-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Security of MSC therapy in very low birth weight preterm babies at risk of developing bronchopulmonary dysplasia | 24 months
  Number of patients with adverse events during the infusion time and during all study; and comorbilities due to preterm birth.
feasibility variable | 24 months
  Number of days of life from birth to administration of the first dose and number of days of life in successive doses.

SECONDARY OUTCOMES:
Incidence of BPD and PH in very low birth weight babies treated with MSC | 24 months
  Status on week 36 of post-menstrual age
Diagnosis and stage of bronchopulmonary dysplasia on week 36 of post-menstrual age according to Jensen | 24 months
  (No BPD/grade 1/grade 2/garde 3)
Exitus on week 36 and 40 of post-menstrual age or at hospital discharge | 24 months
  (Yes/No)
Incidence of comorbidities resulting from prematurity from the time of screening to 40 weeks' EPM, hospital discharge or death. | 24 months
  (sepsis confirmed by blood culture, treated patent ductus arteriosus, non-pharmacological ductal closure, necrotising enterocolitis, isolated bowel perforation, intraventricular haemorrhage ≥ 2, retinopathy ≥ grade 2)
Biomarker analysis (IL-1beta, IL-6, IL8, TGF beta, TNF alfa, GM-CSF, NLRP3, RAGE, HMGB1, VEGF, HGF, GREMLIN1, sVEGFR1, SP-D, SMPD1, SMPD3, IsoPs, IsoFs, NeuroPs, NeuroFs, miRNAs). | 24 months
  biomarkers will be measured in pg/ml
Variations in echocardiographic parameters of pulmonary hypertension (PH) before and after mesenchymal cell therapy. | 24 months
  NO PH (type I less 35%), MILD PH (type I-II between 35-50%) , MODERATE PH (type II between 50-70%) and SEVERE PH ( type II-III, more than 70%)
Changes in modified respirator score during therapy and up to week 36 of port-menstrual age | 24 months
  0 - 13 (min- max value). Higher score means worse outcome.
Changes in Respiratory Severity Score (RSS) during therapy and up to week 36 of port-menstrual age | 24 months
  0-30 (min- max value). Higher score means worse outcome.
Date of hospital discharge and respiratory care at discharge. | 24 months
  Date of hospital discharge and respiratory care at discharge.
Need for supplemental O2 at home discharge and during follow-up (Number if patients that need supplemental O2). | 24 months
  Number if patients that need supplemental O2
Duration of invasive and non-invasive mechanical ventilation. | 24 months
  Duration of invasive and non-invasive mechanical ventilation.
Use of postnatal corticosteroids indicated | 24 months
  For the treatment or prevention of BPD
Respiratory readmission rates. | 24 months
  During the first year
Bayley Neurodevelopmental Scale at 24 months | 24 months
  Evaluation of cognitive developement, languaje developement and motor developement.
Date and cause of death. | 24 months
  Date and cause of death.

CONTACTS AND LOCATIONS:
Overall Officials: María Jesús del Cerro, PhD, Principal Investigator — IRYCIS. Hospital Universitario Ramón y Cajal. Madrid, Spain.
Locations (7):
- Spain (7):
  - Hospital Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Complejo Hospitalario La Coruña, A Coruña
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Carlos Haya, Málaga
  - Hospital Vírgen del Rocío, Seville
  - Hospital Universitario y Politécnico La Fe, Valencia